CLINICAL TRIAL: NCT00748176
Title: The Relationship of Abdominal Circumference and Trunk Length With the Level of Spinal Anesthesia in Obstetric Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Hui-Hsun Huang, Visiting Staff, Department of Anesthesiology, National Taiwan University Hospital
Other Study IDs: 200805027R
Record Dates: First submitted 2008-09-01; First posted 2008-09-08 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Obstetrics for C/S
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — spinal anesthesia with bupivacaine

SUMMARY:
The body shape might have influence on the spinal level. In this research we plan to investigate the relationship of abdominal circumference, trunk length and the level of spinal anesthesia in obstetric patients during Cesarean section.

DETAILED DESCRIPTION:
The level of spinal anesthesia in obstetric patients had been investigated in several studies. Increased cephalad spread of local anesthetics had been demonstrated with increased intra-abdominal pressure, changes in anteroposterior spinal curves and lumbar lordosis. Theoretically the body shape might have contribution to the above factors and might have influence on the spinal level. In this research we plan to investigate the relationship of abdominal circumference, trunk length and the level of spinal anesthesia in obstetric patients during Cesarean section. Only those C/S patients indicated and scheduled for spinal anesthesia will be observed. The spinal anesthesia will be performed as routine practice. This study will not change the clinical plan in any aspect. We will only passively record the abdominal circumference, trunk length and the level of spinal anesthesia and calculate the correlation between them.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric patients for C/S

Exclusion Criteria:

* With major systemic diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Obstetric patients for C/S
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Hsun Huang, Principal Investigator — Department of anesthesiology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan